CLINICAL TRIAL: NCT05673044
Title: Functional Evaluation of Modified Studer and Modified Spiral Orthotopic Ileal Neobladders After Radical Cystectomy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Atef Ali, Assistant lecturer of Urology Assuit University Hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Assuituro
Record Dates: First submitted 2022-12-07; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Orthotopic Neobladders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified Studer ileal neobladder (Experimental): the segment of the iso-peristaltic segment is 8 cm and the total length of the ileum used is 40 cm instead of 60 cm.
  Interventions: Procedure: modified Studer ileal neobladder
- modified spiral ileal neobladder (Experimental): the chimney of the spiral neobladder will be an angled one instead of straight.
  Interventions: Procedure: modified Studer ileal neobladder

INTERVENTIONS:
Procedure: modified Studer ileal neobladder — orthotopic ileal neobladders
  Other Names: modified spiral ileal neobladder

SUMMARY:
Bladder cancer is the most common malignant neoplasm of the urinary system. Neoadjuvant chemotherapy followed by radical cystectomy (RC) is the standard treatment for Muscle invasive bladder cancer.

Studer neobladder is one of the commonly used techniques for orthotopic reconstruction, originally utilizing 60-65 cm of the ileum. However, this leads to formation of a flaccid reservoir.

Nowadays, most techniques use 40-45 cm ileal segment only due to the proven increased reservoir capacity over time. So Moeen et al developed a modified Studer ileal neobladder by using a shorter ileal segment (40 cm only).

Upper urinary tract protection is important in neobladder reconstruction. One of the proposed anti-reflux techniques is using an isoperistaltic limp which was about 20 cm. This segment will be compressed by the elevated intra-abdominal pressure during Valsalva voiding to prevent reflux. However, this length was subjected to multiple reductions in multiple studies. Moeen et al used an 8 cm straight isoperistaltic ileal chimney.

In spiral neobladder the ureters are implanted into the reservoir using a non-refluxing split-cuff nipple technique. It has good functional and urodynamic parameters. Moeen et al added 8 cm as RT sided angled chimney over the neobladder. The ureters were implanted directly in an end to side manner. They assumed that adding this angulation to this short chimney decreases reflux and protect the UUT, without adding time to develop an anti-reflux technique.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with muscle invasive bladder cancer (T2-3N0-1M0).
2. Patients with T1 high grade bladder cancer with failed intravesical immunotherapy.
3. Bladder neck area including the trigone free from cancerous involvement.
4. Patients accepting the operation who are medically fit.

Exclusion Criteria:

1. Patients with serum creatinine ≥ 1.8 mg/dl.
2. Patients with intestinal disorders including previous bowel resections, severe diverticulosis or inflammatory bowel disease.
3. Inability to do perform clean intermittent catheterization (CIC) due to physical or mental impairment.
4. Sphincteric deficiency or urethral stricture disease causing voiding dysfunction.
5. Positive prostatic urethral biopsy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
The assessment of the reservoir capacity | At 3rd month post operative
  Assessment of reservoir capacity by pouch size in urodynamics
The assessment of the reservoir capacity | At 6th month post operative
  Assessment of reservoir capacity by pouch size in urodynamics
The assessment of the reservoir capacity | At 12th month post operative
  Assessment of reservoir capacity by pouch size in urodynamics

CONTACTS AND LOCATIONS:
Overall Officials: Diaa Eldin hameed Sayed, PhD, Study Director — cheif of urological oncology department
Locations (1):
- Assuit university, Asyut, Assuit, Egypt